CLINICAL TRIAL: NCT01337128
Title: Carotid Endarterectomy Versus Carotid Artery Stenting? A Prospective Comparison of Neuropsychological Outcome in Patients With Carotid Stenosis.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Collaborators: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2010/819
Record Dates: First submitted 2011-04-15; First posted 2011-04-18 (Estimated); Last update posted 2021-12-01 (Actual); Status verified 2021-11

CONDITIONS: Carotid Stenosis
MeSH Terms: conditions — Carotid Stenosis | interventions — Endarterectomy, Carotid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Carotid endarterectomy (CEA) (Experimental): Patients with carotid stenosis who are randomly assigned to a carotid endarterectomy.
  Interventions: Procedure: Carotid endarterectomy (CEA); Procedure: Neurocognitive functions; Procedure: Levels of biomarkers; Procedure: Detection of peri-operative embolization; Procedure: Validation results
- Carotid Stenting (CAS) (Experimental): Patients with carotid stenosis who are randomly assigned to a carotid stenting.
  Interventions: Procedure: Carotid stenting (CAS); Procedure: Neurocognitive functions; Procedure: Levels of biomarkers; Procedure: Detection of peri-operative embolization; Procedure: Validation results
- matched control group (No Intervention): Matched control group.

INTERVENTIONS:
Procedure: Carotid endarterectomy (CEA) — Carotid endarterectomy (CEA) will be performed on the patients
  Arms: Carotid endarterectomy (CEA)
Procedure: Carotid stenting (CAS) — Carotid Stenting (CAS) will be performed on these patients.
  Arms: Carotid Stenting (CAS)
Procedure: Neurocognitive functions — Neurocognitive functions will be measured pre-operatively and after 3 weeks, 6 months and 1 year.
  Arms: Carotid Stenting (CAS); Carotid endarterectomy (CEA)
Procedure: Levels of biomarkers — Levels of biomarkers (Protein S100B) will be examined pre- , peri- and post-operatively after 2 hours, 6 hours and 24 hours.
  Arms: Carotid Stenting (CAS); Carotid endarterectomy (CEA)
Procedure: Detection of peri-operative embolization — A Transcranial Doppler Ultrasonography will be used to detect peri-operative embolization.
  Arms: Carotid Stenting (CAS); Carotid endarterectomy (CEA)
Procedure: Validation results — On a subgroup of 20 patients a MRI-scan will be done pre- and post-operatively after 48 hours and 3 weeks.
  Arms: Carotid Stenting (CAS); Carotid endarterectomy (CEA)

SUMMARY:
In this prospective study, patients with carotid stenosis will be randomly assigned to one of the two surgical procedures (carotid endarterectomy (CEA) and carotid stenting (CAS)). Pre- and postoperative neuropsychological functions, levels of several biomarkers and intraoperative embolization load will be examined. In a subgroup of patients, MRI-data will also be gathered. The mix of these data will allow us to answer several questions regarding the absence or presence of preoperative impairments, postoperative changes in cognitive performance and possible differences between CEA and CAS regarding postoperative neuropsychological functions. The use of a matched control group and implementation of a long term follow-up will contribute to the uniqueness of this study. It will meet several flaws of previous studies and will complete the ongoing randomized studies comparing CEA and CAS that are lacking neuropsychological data.

ELIGIBILITY:
Inclusion Criteria:

* Patients with carotid stenosis.

Exclusion Criteria:

* Significant medical conditions which affect neurocognitive functions (e.g. cancer, epilepsy)
* Older than 80 years
* A history of psychiatric or neurological illness
* Severe alcohol of drug abuse
* Coronary artery bypass graft (CABG) less than a year ago.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2011-04 (Actual); Primary Completion 2015-04 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Pre-operative neuropsychological state | pre-operative
  Pen and paper tests will be performed.
Post-operative neuropsychological state (3 weeks) | after 3 weeks
  Pen and paper tests will be performed.
Post-operative neuropsychological state (6 months) | after 6 months
  Pen and paper tests will be performed.
Post-operative neuropsychological state (1 year) | after 1 year
  Pen and paper tests will be performed.

SECONDARY OUTCOMES:
Levels of biomarkers pre-operatively | pre-operatively, intra-operative, after 2 hours, 6 hours and 24 hours
  Levels of biomarkers (protein S100B) will also be examined pre-operatively.
Determination of cardiovascular risks pre-operatively | pre-operatively
  questionnaires
Determination of cardiovascular risks after 3 weeks | after 3 weeks
  questionnaires
Determination of cardiovascular risks after 6 months | after 6 months
  questionnaires
Determination of cardiovascular risks after 1 year | after 1 year
  questionnaires
Clinical neurological examination after 3 weeks | after 3 weeks
Clinical neurological examination after 6 months | after 6 months
Clinical neurological examination after 1 year | after 1 year
Peri-operative embolization | Peri-operative
  A transcranial doppler ultrasonography will be performed.
Validation results | pre- and post-operative after 48 hours and 3 weeks
  MRI-scan will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Frank Vermassen, Ph.D., M.D., Principal Investigator — University Hospital, Ghent; Guy Vingerhoets, Ph.D., Professor, Principal Investigator — University Ghent
Locations (1):
- Ghent University Hospital, Ghent, Belgium